CLINICAL TRIAL: NCT02032069
Title: Pneumoproteins Expression in the Organ Donor
Status: Completed | Type: Observational
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Asmae Belhaj, MD, University Hospital of Mont-Godinne
Other Study IDs: B406201112693
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Primary Graft Dysfunction
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tissues and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NHBD: Non Heart Beating Donors
  Interventions: Other: no intervention
- BDD: Brain death donors
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Primary graft dysfunction, a form of reperfusion pulmonary edema that occurs early after lung transplantation, shares key clinical and pathological features with acute lung injury and its more severe form, the acute respiratory distress syndrome. However, in contrast to acute lung injury/acute respiratory distress syndrome, in which biomarkers in plasma, urine and lung edema fluid have prognostic and pathogenetic value, the role of biomarkers in primary graft dysfunction has been less thoroughly explored. We will try in this study de determine the rule of pneumoproteins in the donor organ on the pulmonary edema in the recipient.

ELIGIBILITY:
Inclusion Criteria:

All the organ donors for lung grafts.

Exclusion Criteria:

none

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Organ donors and lung recipients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of Recipient with primary graft dysfunction | one year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Mont-Godinne, Yvoir, Namur, Belgium